CLINICAL TRIAL: NCT03650868
Title: The Effect of Thoracal Paravertebral Block on Seroma Reduction in Breast Surgery, a Randomised Controlled Trial
Brief Title: The Effect of Thoracal Paravertebral Block on Seroma Reduction in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Alparslan Kus, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KIA 2018/155
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Seroma; Breast Cancer
Keywords: Thoracal Paravertebral Block; Breast Surgery; Seroma Reduction
MeSH Terms: conditions — Seroma; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be applied to control group
- TPVB group (Experimental): Thoracal paravertebral block will be performed with 20cc of 0,25% bupivacaine preoperatively.
  Interventions: Procedure: Thoracal paravertebral block

INTERVENTIONS:
Procedure: Thoracal paravertebral block — Thoracal paravertebral block will be performed before the surgery to the TPVB group.
  Arms: TPVB group

SUMMARY:
Thoracal paravertebral block (TPVB) is a commonly prefferred regional anesthesia technique to provide postoperative analgesia. In addition, the successful use of TPVB is reported for some seroma related pain cases. Postoperative analgesia in breast surgery is a difficult and overworked issue due to etensive surgery and complex innervation of the breast and in addition to this complex mechanisms, seroma accumulation has a negative effect for patients postoperatively. With this study, the investigators aimed to study the effect of TPVB on seroma reduction for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of agge
* ASA I-II
* Undergoing elective breast cancer surgery

Exclusion Criteria:

* obesity (body mass index >35 kg/m2)
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Seroma quantitiy | 24 hour postoperatively.
  Seroma quantitiy of all patients will be recorded after 24 hour postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Kus, Principal Investigator — Kocaeli Üniversitesi Tıp Fakültesi
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No